CLINICAL TRIAL: NCT01891864
Title: A Randomized, Double-blind, Multicenter Study to Demonstrate Equivalent Efficacy and to Compare Safety and Immunogenicity of a Biosimilar Etanercept (GP2015) and Enbrel® in Patients With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Study to Demonstrate Equivalent Efficacy and to Compare Safety of Biosimilar Etanercept (GP2015) and Enbrel
Acronym: EGALITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP15-302
Record Dates: First submitted 2013-06-24; First posted 2013-07-03 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Chronic Stable Plaque Psoriasis
MeSH Terms: interventions — GP2015; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GP2015 Etanercept (Experimental): Solution for subcutaneous injection in pre-filled syringe. The drug is administered in a dose of 50 mg twice weekly for the first 12 weeks and 50 mg once weekly thereafter
  Interventions: Drug: GP2015 Etanercept
- Enbrel ® Etanercept (Active Comparator): Solution for subcutaneous injection in pre-filled syringe. The drug is administered in a dose of 50 mg twice weekly for the first 12 weeks and 50 mg once weekly thereafter
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: GP2015 Etanercept — Sandoz has developed GP2015 Etanercept (Sandoz's code for the drug product containing the active ingredient etanercept) to be biosimilar to Enbrel.
  Other Names: GP2015; Etanercept
  Arms: GP2015 Etanercept
Drug: Enbrel — Enbrel is used as reference product to GP2015.
  Other Names: Etanercept
  Arms: Enbrel ® Etanercept

SUMMARY:
The purpose of this study is to demonstrate equivalent efficacy of GP2015 and Enbrel® in patients with moderate to severe chronic plaque-type psoriasis with respect to PASI 75 response rate at Week 12.

DETAILED DESCRIPTION:
The purpose of this confirmatory safety and efficacy study (GP15-302) was to demonstrate equivalence in efficacy and similarity in safety and immunogenicity of GP2015 and Enbrel (EU-authorized) in patients with moderate to severe chronic plaque-type psoriasis and to evaluate the effects of repeated switching between GP2015 and Enbrel on efficacy, overall safety, and immunogenicity. Since only EU-authorized Enbrel was utilized in this study, the use of the term "Enbrel" throughout this report describes EU-authorized Enbrel only.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age at time of screening
* Chronic plaque-type psoriasis diagnosed for at least 6 months before baseline
* Moderate to severe psoriasis as defined at baseline by:

  * PASI score of 10 or greater and,
  * Investigator´s Global Assessment score of 3 or greater (based on a scale of 0 - 4) and,
  * Body Surface Area affected by plaque-type psoriasis of 10% or greater
* Chronic plaque-type psoriasis patients who have previously received phototherapy or systemic psoriasis therapy at least once or who are candidates for such therapies in the opinion of the investigator.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type
* Drug-induced psoriasis
* Ongoing use of prohibited treatments
* Previous exposure to etanercept
* Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of treatment with etanercept

Other In-/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Gerdes, MD, Principal Investigator — Klinik für Dermatologie, Venerologie und Allergologie Universitätsklinikum Schleswig Holstein, Kiel, Germany
Locations (74):
- Bulgaria (5):
  - Sandoz Investigational Site, Pleven
  - Sandoz Investigational Site, Plovdiv
  - Sandoz Investigational Site 1, Sofia
  - Sandoz Investigational Site 2, Sofia
  - Sandoz Investigational Site 3, Sofia
- Czechia (3):
  - Sandoz Investigational Site, Olomouc
  - Sandoz Investigational Site, Prague
  - Sandoz Investigational Site, Ústí nad Labem
- Estonia (5):
  - Sandoz Investigational Site 1, Tallinn
  - Sandoz Investigational Site 2, Tallinn
  - Sandoz Investigational Site 3, Tallinn
  - Sandoz Investigational Site 1, Tartu
  - Sandoz Investigational Site 2, Tartu
- Germany (7):
  - Sandoz Investigational Site 1, Berlin
  - Sandoz Investigational Site 2, Berlin
  - Sandoz Investigational Site 1, Dresden
  - Sandoz Investigational Site 2, Dresden
  - Sandoz Investigational Site, Kiel
  - Sandoz Investigational Site, Lübeck
  - Sandoz Investigational Site, Munich
- Hungary (4):
  - Sandoz Investigational Site, Budapest
  - Sandoz Investigational Site, Debrecen
  - Sandoz Investigational Site, Gyula
  - Sandoz Investigational Site, Szolnok
- Poland (14):
  - Sandoz Investigational Site, Gdansk
  - Sandoz Investigational Site, Gdynia
  - Sandoz Investigational Site, Katowice
  - Sandoz Investigational Site 1, Krakow
  - Sandoz Investigational Site 2, Krakow
  - Sandoz Investigational Site 1, Lodz
  - Sandoz Investigational Site 2, Lodz
  - Sandoz Investigational Site 3, Lodz
  - Sandoz Investigational Site 4, Lodz
  - Sandoz Investigational Site, Poznan
  - Sandoz Investigational Site, Rzeszów
  - Sandoz Investigational Site, Warsaw
  - Sandoz Investigational Site, Wroclaw
  - Sandoz Investigational Site, Zgierz
- Romania (9):
  - Sandoz Investigational Site, Brasov
  - Sandoz Investigational Site 1, Bucharest
  - Sandoz Investigational Site 2, Bucharest
  - Sandoz Investigational Site 3, Bucharest
  - Sandoz Investigational Site, Cluj-Napoca
  - Sandoz Investigational Site 1, Iași
  - Sandoz Investigational Site 2, Iași
  - Sandoz Investigational Site, Târgu Mureş
  - Sandoz Investigational Site, Timișoara
- Russia (2):
  - Sandoz Investigational Site, Saint Petersburg
  - Sandoz Investigational Site, Smolensk
- Slovakia (8):
  - Sandoz Investigational Site, Banská Bystrica
  - Sandoz Investigational Site, Bojnice
  - Sandoz Investigational Site 1, Bratislava
  - Sandoz Investigational Site 2, Bratislava
  - Sandoz Investigational Site, Kosice-Saka
  - Sandoz Investigational Site, Košice
  - Sandoz Investigational Site, Nitra
  - Sandoz Investigational Site, Svidník
- South Africa (4):
  - Sandoz Investigational Site, Bloemfontein
  - Sandoz Investigational Site, Krugersdorp
  - Sandoz Investigational Site 1, Pretoria
  - Sandoz Investigational Site, Worcester
- Ukraine (8):
  - Sandoz Investigational Site, Dnipropetrovsk
  - Sandoz Investigational Site, Donetsk
  - Sandoz Investigational Site, Kharkiv
  - Sandoz Investigational Site, Kyiv
  - Sandoz Investigational Site, Luhansk
  - Sandoz Investigational Site, Rivne
  - Sandoz Investigational Site, Simferopol
  - Sandoz investigational Site, Zaporizhzhia
- United Kingdom (5):
  - Sandoz Investigational Site, Dundee
  - Sandoz Investigational Site, Leeds
  - Sandoz Investigational Site, London
  - Sandoz Investigational Site, Newcastle upon Tyne
  - Sandoz Investigational Site, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thaci D, Gerdes S, Schulze-Koops H, Allanore Y, Kavanaugh A, Both C, Gattu S, Hachaichi S, Matucci-Cerinic M. Patient-Reported Outcome Measures in Patients with Rheumatoid Arthritis, Psoriasis, or Psoriatic Arthritis Treated with GP2015, an Etanercept Biosimilar: Results from Two Phase III Studies (EGALITY and EQUIRA). Drugs R D. 2025 Jun;25(2):107-115. doi: 10.1007/s40268-025-00507-8. Epub 2025 Apr 25. PMID 40279006

RESULTS

PARTICIPANT FLOW:
Groups:
- GP2015 Etanercept: Solution for subcutaneous injection in pre-filled syringe. The drug is administered in a dose of 50 mg twice weekly for the first 12 weeks and 50 mg once weekly thereafter
  GP2015 Etanercept
- Enbrel ® Etanercept: Solution for subcutaneous injection in pre-filled syringe. The drug is administered in a dose of 50 mg twice weekly for the first 12 weeks and 50 mg once weekly thereafter
  Enbrel ® Etanercept
- GP2015 Etanercept Continued: GP2015 50 mg subcutaneous (s.c.) injection of study drug from week 13 until Week 30 (Treatment Period 2).
  GP2015 50 mg subcutaneous (s.c.) injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2
- Enbrel ® Etanercept Continued: Enbrel ® 50 mg subcutaneous (s.c.) injection of study drug from week 13 until Week 30 (Treatment Period 2) Enbrel ® 50 mg subcutaneous (s.c.) injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
- GP2015 Etanercept Switched: GP2015/Enbrel ® 50 mg subcutaneous (s.c.) injection of study drug until Week 30. Three periods of 6 weeks alternating between Enbrel/GP2015/Enbrel (Treatment Period 2).
  Enbrel ® 50 mg subcutaneous (s.c.) injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
- Enbrel ® Etanercept Switched: Enbrel ®/GP2015 50 mg subcutaneous (s.c.) injection of study drug until Week 30. Three periods of 6 weeks alternating between GP2015/Enbrel/GP2015 (Treatment Period 2).
  GP2015 50 mg subcutaneous (s.c.) injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
Period: Treatment Period 1
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept | GP2015 Etanercept Continued | Enbrel ® Etanercept Continued | GP2015 Etanercept Switched | Enbrel ® Etanercept Switched
Started | 264 | 267 | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period) | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period) | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period) | 0 (Treatment arm applicable only in Treatment Period 2 and Extension Period)
Completed | 256 (6 patients discontinued after completion of Treatment Period 1 and did NOT start Treatment Period 2) | 255 (8 patients discontinued after completion of Treatment Period 1 and did NOT start Treatment Period 2) | 0 | 0 | 0 | 0
Not Completed | 8 | 12 | 0 | 0 | 0 | 0
Not completed — Protocol Violation / IMP non-compliance | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event, Serious, Fatal | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event / Injection Site Reaction | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept | GP2015 Etanercept Continued | Enbrel ® Etanercept Continued | GP2015 Etanercept Switched | Enbrel ® Etanercept Switched
Started | 0 (Treatment arm applicable for Treatment Period 1 only (patients re-randomized in Treatment Period 2)) | 0 (Treatment arm applicable for Treatment Period 1 only (patients re-randomized in Treatment Period 2)) | 150 (Part of the patients re-randomized from "GP2015 Etanercept" treatment arm in Treatment Period 1) | 151 (Part of the patients re-randomized from "Enbrel ® Etanercept" treatment arm in Treatment Period 1) | 100 (Part of the patients re-randomized from "GP2015 Etanercept" treatment arm in Treatment Period 1) | 96 (Part of the patients re-randomized from "Enbrel ® Etanercept" treatment arm in Treatment Period 1)
Completed | 0 | 0 | 143 | 142 | 96 | 91
Not Completed | 0 | 0 | 7 | 9 | 4 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Site Termination | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0 | 4
Not completed — Termination of Site | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 4 | 1 | 1
Period: Extension Period
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept | GP2015 Etanercept Continued | Enbrel ® Etanercept Continued | GP2015 Etanercept Switched | Enbrel ® Etanercept Switched
Started | 0 | 0 | 140 (2 patients withdrew consent 1 patient lost to FU between Treatment Period 2 and the Extension period) | 142 | 95 (1 patient discontinued between Treatment Period 2 and Extension Period due to lack of efficacy) | 90 (1 patient discontinued between Treatment Period 2 and Extension Period due to an adverse event)
Completed | 0 | 0 | 132 | 137 | 88 | 90
Not Completed | 0 | 0 | 8 | 5 | 7 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized in GP15-302 study
Groups:
- Total: Total of all reporting groups
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept | Total
Number analyzed (Participants) | 264 | 267 | 531
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 254 | 249 | 503
  >=65 years | 10 | 18 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (12.29) | 42.7 (12.86) | 42.4 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 95 | 202
  Male | 157 | 172 | 329
Region of Enrollment [Number; unit: participants]
  Czech Republic | 25 | 16 | 41
  Russian Federation | 9 | 8 | 17
  Romania | 9 | 24 | 33
  Hungary | 9 | 12 | 21
  Ukraine | 19 | 23 | 42
  Poland | 96 | 94 | 190
  South Africa | 4 | 1 | 5
  United Kingdom | 10 | 4 | 14
  Slovakia | 17 | 20 | 37
  Bulgaria | 13 | 8 | 21
  Germany | 12 | 17 | 29
  Estonia | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: PASI 75 Response Rate at Week 12 - GP2015 Etanercept vs. Enbrel ® Etanercept
Description: The 95% CI for the Psoriasis Area and Severity Index (PASI) 75 response rate differences at Week12 between GP2015 Etanercept and Enbrel ® Etanercept. PASI 75 response: patients who achieved ≥ 75% improvement (reduction) in PASI score compared to baseline were defined as PASI 75 responders. PASI scores can range from 0, corresponding to no signs of psoriasis up to theoretic maximum of 72.0, which means a higher PASI score reflects a higher psoriasis activity.
Time Frame: Week 12
Population: The analysis of the primary outcome measure was based on the per-protocol set (PPS) consisting of patients who completed study until 12 weeks without any major protocol deviation.
Measure: Number; unit: % of patients achieving PASI75 response
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept
Number analyzed (Participants) | 239 | 241
% of patients achieving PASI75 response | 73.4 | 75.7
Statistical Analysis 1: Comparison: GP2015 Etanercept vs Enbrel ® Etanercept; PASI 75 response rate (proportion of patients showing at least a 75% improvement in PASI) after the first 12 weeks of treatment (Treatment Period 1) was the primary endpoint to assess equivalence between GP2015 and Enbrel®. Therapeutic equivalence in terms of PASI75 could be concluded if the exact 95% confidence interval for the difference in the PASI75 rates is completely contained within the interval [-18%; 18%]. A logistic regression model was to be employed; Test type: Non-Inferiority or Equivalence — The equivalence margin for the comparison of GP2015 with Enbrel with respect to PASI 75 response at Week 12 was based on response rates reported in two pivotal placebo controlled trials (Leonardi et al 2003; Papp et al 2005). Based on the observed effect size of 45-46%, an equivalence margin of 18% was chosen so that at least 60% of the treatment effect seen for Enbrel was maintained. A response rate of 49% was assumed for the comparator treatment Enbrel; Risk Difference (RD) = -2.3, 95% CI 2-sided [-9.85 to 5.3]

2. Secondary Outcome: Percent Change From Baseline in PASI Score up to Week 12
Description: The key secondary efficacy endpoint was the % change from baseline in PASI score up to Week 12. PASI scores can range from 0, corresponding to no signs of psoriasis up to theoretic maximum of 72.0, which means a higher PASI score reflects a higher psoriasis activity. Two approaches (longitudinal approach applying a Mixed Model Repeated Measures and Averaged Treatment Effect approach applying an ANCOVA model) were employed in order to calculate 2-sided 95% confidence intervals (CI) for the difference between the treatment groups.
Time Frame: 12 weeks
Population: The analysis was based on the per-protocol set (PPS) consisting of patients who completed study until 12 weeks without any major protocol deviation.
Measure: Least Squares Mean (Standard Error); unit: percentage difference
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept
Number analyzed (Participants) | 239 | 241
percentage difference | -56.11 (1.0578) | -55.48 (1.0511)
Statistical Analysis 1: Comparison: GP2015 Etanercept vs Enbrel ® Etanercept; Test type: Non-Inferiority or Equivalence — A MMRM (Mixed Model Repeated Method) was performed on the percentage change from baseline in PASI score from baseline to Week 12. Therapeutic equivalence in terms of the % change from baseline in PASI score was to be determined if the 95% CI for the difference between GP2015 and Enbrel was contained within the interval [-15%; 15%]; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-3.474 to 2.204]
Statistical Analysis 2: Comparison: GP2015 Etanercept vs Enbrel ® Etanercept; Test type: Non-Inferiority or Equivalence — The mean averaged treatment effect (ATE) of percent change from baseline in PASI score up to week 12 was derived for each patient and analyzed using an ANCOVA approach. Therapeutic equivalence in terms of the % change from baseline in PASI score was to be determined if the 95% CI for the difference between GP2015 and Enbrel was contained within the interval [-15%; 15%]; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-3.61 to 1.845]

3. Secondary Outcome: PASI 50, 75 and 90 Response Rates
Description: Percentage of patients achieving Psoriasis Area and Severity Index (PASI) 50, PASI 75, and PASI 90 responses at Week 12. PASI 50 response: patients who achieved ≥ 50% improvement (reduction) in PASI score compared to baseline were defined as PASI 50 responders .PASI 90 response: patients who achieved ≥ 90% improvement (reduction) in PASI score compared to baseline were defined as PASI 90 responders .
Time Frame: Week12
Population: The analysis of this secondary outcome measure was based on the per-protocol set (PPS) consisting of patients who completed study until 12 weeks without any major protocol deviation.
Measure: Number; unit: percentage of patients
Arm/Group | GP2015 Etanercept | Enbrel ® Etanercept
Number analyzed (Participants) | 239 | 241
percentage of patients
  % of patients achieving PASI50 response at Week 12 | 99.2 | 97.9
  % of patients achieving PASI75 response at Week 12 | 73.4 | 75.7
  % of patients achieving PASI90 response at Week 12 | 39.2 | 34.1

4. Secondary Outcome: Injection Site Reactions
Description: Percentage of patients with injection site reactions up to Week 52
Time Frame: Week52
Population: The analysis was performed on safety set including all patients who took at least 1 dose of study treatment
Measure: Number; unit: percentage of patients with ISRs
Groups:
- GP2015 Etanercept Continued: GP2015 Etanercept (s.c.) injection administered in a dose of 50 mg twice weekly for the first 12 weeks.
  GP2015 Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug from week 13 until Week 30 (Treatment Period 2).
  GP2015 Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
- Enbrel ® Etanercept Switched: Enbrel ® Etanercept (s.c.) injection administered in a dose of 50 mg twice weekly for the first 12 weeks.
  Enbrel ® Etanercept /GP2015 Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug until Week 30. Three periods of 6 weeks alternating between GP2015/Enbrel/GP2015 (Treatment Period 2).
  GP2015 Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
- GP2015 Etanercept Switched: GP2015 Etanercept (s.c.) injection administered in a dose of 50 mg twice weekly for the first 12 weeks.
  GP2015 Etanercept /Enbrel ® Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug until Week 30. Three periods of 6 weeks alternating between Enbrel/GP2015/Enbrel (Treatment Period 2).
  Enbrel ® Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
- Enbrel ® Etanercept Continued: Enbrel ® Etanercept (s.c.) injection administered in a dose of 50 mg twice weekly for the first 12 weeks.
  Enbrel ® Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug from week 13 until Week 30 (Treatment Period 2).
  Enbrel ® Etanercept 50 mg subcutaneous (s.c.) weekly injection of study drug from week 31 until Week 52 (Extension Period) in patients who had completed Treatment Period 2.
Arm/Group | GP2015 Etanercept Continued | Enbrel ® Etanercept Switched | GP2015 Etanercept Switched | Enbrel ® Etanercept Continued
Number analyzed (Participants) | 164 | 96 | 100 | 171
percentage of patients with ISRs | 8.5 | 16.7 | 9.0 | 15.8

5. Secondary Outcome: Immunogenicity: Measurement of Rate of ADA Formations Against GP2015 Etanercept and Enbrel ® Etanercept
Description: Immunogenicity was analyzed by the percentage of patients with positive anti-drug antibodies (ADA) to either GP2015 Etanercept or Enbrel ® up to Week 52.
Time Frame: Week 52
Population: The analysis was performed on immunogenicity set consisting of patients who provided data for ADA assessment of etanercept at baseline visit.
Measure: Number; unit: percentage patients with positive ADA
Arm/Group | GP2015 Etanercept Continued | Enbrel ® Etanercept Switched | GP2015 Etanercept Switched | Enbrel ® Etanercept Continued
Number analyzed (Participants) | 140 | 90 | 95 | 142
percentage patients with positive ADA | 0 | 1.1 | 0 | 3.5

ADVERSE EVENTS:
Time Frame: Adverse events are reported until the end of the study (week 52).
Arm/Group | GP2015 Etanercept Continued | Enbrel ® Etanercept Switched | GP2015 Etanercept Switched | Enbrel ® Etanercept Continued
Serious Adverse Events (participants affected / at risk) | 7/164 | 6/96 | 6/100 | 7/171
Other Adverse Events (participants affected / at risk) | 97/164 | 57/96 | 60/100 | 94/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP2015 Etanercept Continued (N=164) | Enbrel ® Etanercept Switched (N=96) | GP2015 Etanercept Switched (N=100) | Enbrel ® Etanercept Continued (N=171)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milk allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Fatal event
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acid-base balance disorder mixed (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP2015 Etanercept Continued (N=164) | Enbrel ® Etanercept Switched (N=96) | GP2015 Etanercept Switched (N=100) | Enbrel ® Etanercept Continued (N=171)
Hypertenson (Vascular disorders) | 5 (5) | 2 (2) | 3 (3) | 7 (8)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 6 (6) | 2 (2) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 6 (6) | 0 (0) | 3 (3) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (7) | 4 (5) | 8 (8)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Schiatica (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (5) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (9) | 3 (4) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (26) | 10 (15) | 14 (16) | 17 (22)
Pharyngitis (Infections and infestations) | 7 (9) | 3 (4) | 5 (5) | 10 (11)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6) | 8 (12) | 4 (6) | 6 (7)
Respiratory tract infection viral (Infections and infestations) | 4 (6) | 1 (1) | 4 (4) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3) | 1 (2) | 5 (9)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 3 (4)
Rhinitis (Infections and infestations) | 2 (2) | 3 (4) | 1 (1) | 4 (5)
Tonsillitis (Infections and infestations) | 5 (6) | 1 (1) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Cystitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty days prior to submitting/presenting manuscript or other materials relating to the study a copy should be provided to Sandoz and Sandoz has sixty days to review and comment. Sandoz has the right to require amendments to any such proposed presentation or publication on reasonable grounds. Sandoz may require any proposed publication or presentation to be delayed for up to four months to enable a patent application to be prepared and filed.